CLINICAL TRIAL: NCT02594670
Title: Acupuncture Based on Different Acupoints Combination for Insomnia: a Randomized Controlled Trial
Brief Title: Acupuncture for Insomnia: a Randomized Controlled Trial
Acronym: AI-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other)
Collaborators: University of British Columbia (Other); Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014CB543102-1
Record Dates: First submitted 2014-09-30; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-03

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: acupoints; insomnia; acupuncture; randomized controlled trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DU20 and HT7 combination (Experimental): combination of two acupoints based on location and Heart meridian, including Baihui (DU20) and Shenmen(HT7).
  Interventions: Other: DU20 and HT7 combination
- DU20 and SP6 combination (Other): combination of two acupoints based on location and Spleen meridian, including Baihui (DU20) and Sanyinjiao(SP6).
  Interventions: Other: DU20 and SP6 combination
- DU20 and SA combination (Sham Comparator): combination of local acupoint Baihui (DU20) and a sham acupoint (SA) not belonging to any regular meridian or acupoint.
  Interventions: Other: DU20 and SA combination

INTERVENTIONS:
Other: DU20 and HT7 combination — acupoints combination includes Baihui (DU20) and Shenmen(HT7),which was considered as the optimal clinical efficay among various combinations of acupoints.
  Arms: DU20 and HT7 combination
Other: DU20 and SP6 combination — acupoints combination of Baihui (DU20) and Sanyinjiao (SP6), which should have some clinical efficay among various combinations of acupoints.
  Arms: DU20 and SP6 combination
Other: DU20 and SA combination — Combination of Baihui (DU20) and a Sham acupoint (SA), which should have least clinical efficacy among these three types of acupoints combinations.
  Arms: DU20 and SA combination

SUMMARY:
Selecting different acupoints as an combination of acupoints is a key factor to clinical efficacy of acupuncture. Different combinations of acupoints will generate different clinical efficacy. So,the purpose of this study is to determine the different clinical efficacy among three types of combinations of acupoints in the treatment of primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as insomnia based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition,2013, American psychiatric association
* PSQI score >7
* AIS score ≥6
* SDS ≤60
* SAS ≤60
* Age between 18 and 65 years old
* Not involved in other clinical trial in the lasted 6 months before screening
* Have the ability to write the informed consent.

Exclusion Criteria:

* Breathing-related sleep disorders
* Circadian rhythm sleep-wake disorders
* Medication-induced sleep disorder
* Substance induced sleep disorders,such as alcohol, coffee, strong tea
* Secondary insomnia caused by systemic diseases or caused by external environment disturbance
* Pregnant or lactating women
* Combined with serious cardiovascular, lung, liver, kidney, hematopoietic system, and mental diseases
* Advanced malignant tumor or other serious debilitating diseases
* Location of acupoints combined with infection and bleeding
* Declined to acupuncture
* Couldn't provide the written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index (PSQI) | 4 weeks

SECONDARY OUTCOMES:
Athens Insomnia Scale (AIS) | 4 weeks and 8 weeks
Short Form 36-item Health Survey(SF-36) | 4 weeks and 8 weeks
Self-anxiety scale (SAS) | 4 weeks and 8 weeks
Self-depression scale (SDS) | 4 weeks and 8 weeks

OTHER OUTCOMES:
safety evaluation will summarize the incidence of adverse events，including itching and redness of local acupoints. | 4 weeks
adherence of acupuncture | 4 weeks
  adherence to the treatment (adherence rate)will be calculated using formula: Adherence Rate = Number of Treatment Conducted/ Number of Treatment Planned

CONTACTS AND LOCATIONS:
Overall Officials: Zenghui Yue, Study Chair — Hunan University of Chinese Medicine
Locations (3):
- China (3):
  - Second Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - First Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - Hengyang hospital of Hunan University of Chinese Medicine, Hengyang, Hunan